CLINICAL TRIAL: NCT07269652
Title: HappyOrNot® Smileys and the Visual Analogue Scale (VAS) in the Assessment of Urinary Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seinajoki Central Hospital (Other)
Collaborators: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Mika Raitanen, M.D., Ph.D, Associate Professor, Tampere University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R22025
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Prostate Hyperplasia
Keywords: urinary symptom questionnaries; Visual analogy scale
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Pain Measurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VAS and NoH and urinary symptoms (Experimental): Participants with prostate hyperplasia
  Interventions: Diagnostic Test: Visual analogue scale and HappyorNot smileys

INTERVENTIONS:
Diagnostic Test: Visual analogue scale and HappyorNot smileys — VAS and HoN has not been studied before
  Other Names: Symptom questionnary

SUMMARY:
INTRODUCTION A simple and repeatable test would be valuable for assessing the severity and impact of urinary symptoms. Visual Analogue Scale (VAS) is a 10 cm line where a participant put a mark in place that describes best his satisfaction with woiding. VAS has been shown to correlate with flowmetry and International Prostate Symptom Score (IPSS). VAS is still a number and may not reflect participants satisfaction. HappyorNot smileys (HoN) (emoji faces) are used to measure customer satisfaction by pressing one of four emoji smilyes. Two of these are happy and two and unhappy.

OBJECTIVE:

- To study the use of VAS and HoN in assessing urinary symptoms in men.

MATERIALS AND METHODS:

* 100 men referred to urology outpatient clinic in Tampere University Hospital or Seinäjoki Central Hospital due to urinary symptoms caused by benign Prostate Hyperplasia (BPH)
* Participants are asked to fill VAS and HoN and results are correlated with traditional symptom questionnaires and peak urinary flow and post-void residual volume.

DETAILED DESCRIPTION:
Introduction

Several validated questionnaires have been developed to assess the severity and impact of urinary symptoms, using different sets of questions and scoring methods. Although these tests can provide an accurate assessment of patients' symptoms and the bother caused by them, their clinical usability is limited. Some patients have difficulty completing and understanding the questionnaires without assistance. In addition, analysing multi-item questionnaires based on numerical values is time-consuming, and their repeatability in clinical practice is questionable.

A simple, easy-to-use, and easily repeatable test would be valuable for assessing the severity and impact of urinary symptoms. One possibility is the Visual Analogue Scale (VAS), where the patient evaluates symptom severity or bother on a 10-cm line, with one end representing no symptoms/no bother and the other end representing the worst possible symptom/bother.

VAS scales have been used successfully for many years, particularly in pain assessment. For example, in urogynecological conditions, VAS has been shown to be a functional and reproducible tool compared with validated questionnaires. However, some negative findings have also been reported regarding its use in assessing urinary incontinence in women.

The use of VAS for evaluating lower urinary tract symptoms in men has been studied. The study compared VAS with the seven symptoms assessed by the IPSS questionnaire and found a good correlation. VAS compared with IPSS has also been studied in prostate cancer patients undergoing radiation therapy, where VAS performed even better than IPSS in measuring quality of life. The clinical validation of VAS for urinary symptoms has been reported in one study of 1,000 men, showing good correlation with both IPSS and uroflowmetry. In our own pilot study, VAS correlated well with the EPIC-26 questionnaire when assessing post-prostatectomy urinary symptoms.

Another very simple method for assessing urinary symptoms, their bother level, and response to medical or surgical treatment could be the use of HappyOrNot® smileys (emoji faces). These have long been used to measure customer satisfaction with a single button press. They provide an easy overview of customer satisfaction and have even been shown to increase it, which is why they are commonly seen at service points. However, no studies exist on the use of these smileys to evaluate the impact of medical treatments on patients' symptom experiences.

Objective and Study Material

Some pilot studies have assessed the use of VAS in evaluating urinary symptoms in men, but no large validation studies exist. HappyOrNot® smileys have not previously been used for medical purposes to assess symptom severity or treatment response. The aims of this study is:

To validate the use of HappyOrNot® smileys and the VAS scale in assessing urinary symptoms in men referred to the urology outpatient clinic, using the DAN-PSS questionnaire as the reference. In addition, to investigate the association between HappyOrNot®/VAS results and objective measures of urinary symptom severity, such as peak urinary flow and post-void residual volume.

In the first phase, men referred to the urology outpatient clinic at Tampere University Hospital (TAYS) or Seinäjoki Central Hospital due to urinary symptoms likely caused by benign prostatic hyperplasia will be recruited. This pilot aims to test the correlation of HappyOrNot® and VAS results with the widely used DAN-PSS questionnaire. A total of 100 suitable men will be recruited.

Study Procedure Patients will receive, in addition to the standard appointment letter, the HappyOrNot® smileys, the VAS scale, the DAN-PSS questionnaire, and the study information and consent form. Patients bring the completed forms to their appointment. The consent form is reviewed and signed during the visit. If the patient has questions, the clinician answers them. If the patient forgot the forms, they may complete them before the appointment.

The following data will be collected: HappyOrNot® result, VAS scores, DAN-PSS results, age, prostate size, uroflowmetry (voided volume and peak flow), and post-void residual volume.

Statistical Analysis Spearman correlation will be used to compare HappyOrNot® and VAS results with the clinical questionnaire. Receiver operating characteristic (ROC) analysis will be used to evaluate the classification ability of HappyOrNot® and VAS in determining urinary symptom severity compared with validated questionnaires.

Power Calculation Based on pilot data, where a correlation of 0.722 was found between VAS and EPIC-26 in 200 patients, the power calculation was performed. With a power of 0.8 and significance level of 0.05, only 14 patients would be required. However, since this is a validation study requiring ROC analyses and considering possible dropouts, the sample size for Phase 1 is set to 100.

Study Registry

A study registry will be established and maintained on a secure Tampere University Hosptital (TAYS) hard drive in the Lokero database. Access is restricted to study researchers.

Data will be collected at each centre using the TAYS-maintained RedCap system. Centers are responsible for secure storage and destruction of paper forms (consent and questionnaires). Data transferred to RedCap will be pseudonymised. The system assigns each patient a study number. All analyses use this study number. Results will be published at group level so that individual participants cannot be identified.

A list linking personal identifiers with study numbers will be stored for 25 years at each centre and is accessible only to that centre's researchers and the principal investigators.

Timeline Study started in autumn 2022 and patient recruitment was completed in 2025. Data will be analysed in the early of 2026. Study focuses on evaluating the correlation between HappyOrNot®, VAS, and DAN-PSS.

All results will be published in international peer-reviewed journals. Ethical Considerations A fast, reliable, and easy-to-use tool is needed for assessing urinary symptoms in clinical care. VAS is already a validated and simple method for evaluating pain and may be useful for other symptoms as well. No prior research exists on using HappyOrNot® smileys for assessing symptoms or treatment outcomes.

In this study, patients undergo no procedures outside normal clinical practice. The only additional burden is completing the HappyOrNot® and VAS assessments alongside existing questionnaires. All study-related assessments occur during routine care, so the study does not add workload. Participation is voluntary, requires informed consent, and does not affect treatment. Patients may withdraw at any time.

The study protocol has been approved by TAYS Ethics Committee in June 2022 (ref number R22025). HappyOrNot® -Company has provided written permission for the research use of their smileys.

ELIGIBILITY:
Inclusion Criteria:

* all men having urinary symptoms due to prostate hyperplasia

Exclusion Criteria:

* not signing informed consent

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
HappyorNot smileys and Visual Analogue Scale in the assesment of urinary symptoms | From enrollment to the end of outpatient clinic visit
  HappyOrNot® smileys (four faces of which two represent different degrees of happyness and two different degree of unhappyness) and the Visual Analog Scale (0-10 cm, 0 cm meaning total unsatisfaction and 10 cm meanning total satisfaction) assessing urinary symptoms in men referred to the urology outpatient clinic, using traditional questionnaire as the reference. In addition, to investigate the association between HappyOrNot®/VAS results and objective measures of urinary symptom severity, such as peak urinary flow and post-void residual volume.

CONTACTS AND LOCATIONS:
Overall Officials: Mika Petri Raitanen, M.D., Ph.D., Associate Prof, Study Director — Seinajoki Central Hospital
Locations (1):
- Seinajoki Central Hospital, Seinäjoki, Finland

IPD SHARING:
Plan to Share IPD: Yes
SPSS data
Supporting Information: Study Protocol, CSR
Time Frame: from March 2026 to December 2026